CLINICAL TRIAL: NCT01488435
Title: Efficacy and Tolerance of a Follow-On Formula Fed to Children From 36-48 Months of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Shanghai Children's Medical Center (Other); Shanghai, China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6012
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Acute Respiratory Infection; Diarrheal Disease
MeSH Terms: interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cow's Milk (Placebo Comparator): Powdered whole cow's milk
  Interventions: Dietary Supplement: Cow's milk
- Follow-On Formula (Experimental): Powdered Follow-On Formula with added long-chain Polyunsaturated fatty acid, prebiotics, and polysaccharide
  Interventions: Dietary Supplement: Follow-On Formula

INTERVENTIONS:
Dietary Supplement: Cow's milk — Powdered whole cow's milk
  Arms: Cow's Milk
Dietary Supplement: Follow-On Formula — Powdered Follow-On Formula with added long-chain Polyunsaturated fatty acid, prebiotics, and polysaccharide
  Arms: Follow-On Formula

SUMMARY:
The purpose is to determine if the consumption of study product has an effect on acute respiratory infections and/or diarrheal disease.

ELIGIBILITY:
Inclusion Criteria:

* Child 36-48 months of age
* Child is currently attending a daycare and has attended for 6 months or less
* Has consumed cow's milk or a cow's milk-based beverage during the 48 hours prior to randomization
* Signed informed consent

Exclusion Criteria:

* Child who received any food product or supplement containing probiotics or prebiotics in the 15 days prior to randomization
* Child with allergy to gluten or serious concurrent illness that will interfere in the general management of the child
* Child with diarrhea or acute respiratory infection during the 48 hours prior to randomization
* Child's z-score of weight for height < -3 according to World Health Organization criteria

Ages: 36 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Acute respiratory infections and diarrheal disease | 28 weeks

SECONDARY OUTCOMES:
Allergic manifestations | 28 weeks
Systemic antibiotic use | 28 weeks
Duration of acute respiratory infection and diarrheal disease | 28 weeks
Changes in stool patterns | Baseline and 28 weeks
Fecal immune markers | Baseline and 28 weeks
Serum Ferritin status | Baseline and 28 weeks
Incidence of stool parasites | Baseline and 28 weeks
Growth | 28 weeks
Adverse events | 28 weeks
  The incidence of any adverse event for each participant
Acceptance of study product | 28 weeks
  Acceptance of study product based on quantity consumed.
Serum immune markers | Baseline and 28 weeks
Serum zinc status | Baseline and 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xingming Jin, M.D., Principal Investigator — Professor of Development and Behavioral Pediatrics, Shanghai Children Medical Center
Locations (1):
- Shi-ji-xing Child Care Center, Jin Dong District, Jinhua, Zhejiang, China

REFERENCES:
- [Derived] Li F, Jin X, Liu B, Zhuang W, Scalabrin D. Follow-up formula consumption in 3- to 4-year-olds and respiratory infections: an RCT. Pediatrics. 2014 Jun;133(6):e1533-40. doi: 10.1542/peds.2013-3598. Epub 2014 May 19. PMID 24843061